CLINICAL TRIAL: NCT02574520
Title: A Placebo-controlled (Part 1) or Active-controlled (Part 2) Trial of SABER® -Bupivacaine for the Management of Postoperative Pain Following Laparoscopic Cholecystectomy (PERSIST)
Brief Title: Trial of Extended Release Bupivacaine for Pain Relief After Surgery
Acronym: PERSIST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Durect (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C803-028
Record Dates: First submitted 2015-10-09; First posted 2015-10-14 (Estimated); Results first posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-06

CONDITIONS: Post Operative Pain
Keywords: Post-operative pain; non-opioid analgesic; opioid reduction; laparoscopic cholecystectomy; laparoscopic surgery; bupivacaine; extended release; locally acting analgesic
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Placebo Comparator): SABER-Bupivacaine and Saline Placebo
  Interventions: Drug: SABER-Bupivacaine (Part 1); Drug: Saline Placebo
- Part 2 (Active Comparator): SABER-Bupivacaine and Bupivacaine HCl
  Interventions: Drug: SABER-Bupivacaine (Part 2); Drug: Bupivacaine HCl

INTERVENTIONS:
Drug: SABER-Bupivacaine (Part 1) — 5 ml once at end of surgery
  Other Names: POSIMIR® bupivacaine solution
  Arms: Part 1
Drug: SABER-Bupivacaine (Part 2) — 5 ml once at end of surgery
  Other Names: POSIMIR® bupivacaine solution
  Arms: Part 2
Drug: Saline Placebo — 5 ml once at end of surgery
  Other Names: placebo
  Arms: Part 1
Drug: Bupivacaine HCl — 0.5%, 15 ml, once at end of surgery
  Arms: Part 2

SUMMARY:
This is a research study of SABER® -Bupivacaine, an experimental medication designed to reduce pain for up to 3 days after surgery. Given once by the surgeon at the end of surgery, SABER® - Bupivacaine delivers a locally-acting pain reliever directly to the surgical wound.

The purpose of this study is to measure how well it works in reducing pain after laparoscopic cholecystectomy (surgery to remove the gall bladder) and to investigate the safety of SABER®-Bupivacaine (its side effects).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective outpatient laparoscopic cholecystectomy using a conventional 4-port laparoscopic procedure.
* Must be able and willing to provide written informed consent, complete trial-related procedures, and communicate with the trial staff.
* Males and females 18 years of age or older.
* ASA Class I, II, or III.
* Patients of child-bearing potential must agree to use a medically acceptable method of contraception to prevent pregnancy for the duration of their participation in the trial.
* Must be living close enough to the investigative site to attend the four scheduled follow-up clinic visits.

Exclusion Criteria:

* Pregnant or nursing females.
* Patients with absolute or relative contraindications to laparoscopic cholecystectomy.
* Patients with prior midline abdominal surgery who are at risk for adhesions that may complicate laparoscopic cholecystectomy and/or accurate pain assessments.
* Patients requiring emergency surgery or urgent surgery (fewer than 5 days between screening and surgery).
* Patients with a pre-planned overnight stay or pre-planned hospital admission.
* Patients scheduled for single incision, mini trocars, natural orifice transluminal endoscopic surgery (NOTES), robotic laparoscopic procedures, or any procedure (other than cholangiograms and minimal adhesiolysis) in addition to laparoscopic cholecystectomy.
* Patients with known hypersensitivity to amide local anesthetics such as bupivacaine.
* Patients with acute pain that is not due to cholecystitis.
* Patients with a history of chronic pain unrelated to gallbladder disease.
* Patients with ongoing depression or psychosis.
* Patients undergoing long-term treatment with opioids or other analgesics, including acetaminophen, NSAIDs, anticonvulsants (gabapentin or pregabalin), and antidepressants (SSRIs, SNRIs, and tricyclics), but not including daily low-dose aspirin.
* Patients who are being treated chronically with systemic corticosteroids or who will require peri-operative corticosteroids because of adrenal insufficiency (inhalational or topical corticosteroids are permitted).
* Patients who may be unsuitable for opioid administration (such as sensitivity [e.g., history of severe nausea and vomiting] hypersensitivity, known history of abuse or addiction, or unwillingness to take prescribed rescue opioids).
* Use of anticoagulants and antiplatelet drugs (with exception of low dose aspirin) in the 1 week prior to surgery.
* Patients who are incapable of operating the electronic diary.
* Patients participating in any other trial with an investigational drug or device concurrently or less than 30 days prior to surgery for this trial.
* Patients who, in the Investigator's opinion, should not participate in the trial or may not be capable of following the trial procedures for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dave Ellis, MD, Study Director — Durect
Locations (21):
- United States (21):
  - Durect Study Site 04, Florence, Alabama
  - Durect Study Site 03, Sheffield, Alabama
  - DURECT Study Site 24, Arcadia, California
  - Durect Study Site 15, Fontana, California
  - Durect Study Site 02, Laguna Hills, California
  - Durect Study Site 18, Laguna Hills, California
  - Durect Study Site 22, Pensacola, Florida
  - Durect Study Site 12, Indianapolis, Indiana
  - Durect Study Site 21, Royal Oak, Michigan
  - Durect Study Site 17, Jackson, Mississippi
  - Durect Study Site 16, Las Vegas, Nevada
  - Durect Study Site 20, Las Vegas, Nevada
  - Durect Study Site 05, Stony Brook, New York
  - Durect Study Site 13, Durham, North Carolina
  - Durect Study Site 09, Cleveland, Ohio
  - Durect Study Site 11, Cleveland, Ohio
  - Durect Study Site 07, Cleveland, Ohio
  - Durect Study Site 14, Philadelphia, Pennsylvania
  - Durect Study Site 08, Houston, Texas
  - DURECT Study Site 01, Houston, Texas
  - Durect Study Site 23, Plano, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 22 sites in the US. First subject was randomized on 17 November 2015. Study completion date was on 16 Aug 2017.
Groups:
- Saline Placebo (Part 1); SABER-Bupivacaine (Part 2): 5 ml once at end of surgery
- Bupivacaine HCL (Part 2): 0.5%, 15 ml, once at end of surgery
Period: Overall Study
Arm/Group | SABER-Bupivacaine (Part 1) | Saline Placebo (Part 1) | SABER-Bupivacaine (Part 2) | Bupivacaine HCL (Part 2)
Started (Subjects randomized) | 48 | 46 | 153 | 152
Dosed (ITT subjects who are randomized and dosed. One subject in Part 1 was randomized to receive SABER-Bupivacaine but was treated with Saline Placebo (the safety population includes subjects as randomized).) | 46 | 46 | 148 | 148
Completed | 46 | 46 | 148 | 144
Not Completed | 2 | 0 | 5 | 8
Not completed — Not dosed | 2 | 0 | 5 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All Enrolled Subjects (ITT population)
Groups:
- Total: Total of all reporting groups
Arm/Group | SABER-Bupivacaine (Part 1) | Saline Placebo (Part 1) | SABER-Bupivacaine (Part 2) | Bupivacaine HCL (Part 2) | Total
Number analyzed (Participants) | 48 | 46 | 153 | 152 | 399
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (14.2) | 41.8 (12.8) | 45.5 (13.5) | 44.7 (13.9) | 44.8 (13.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 29 | 115 | 117 | 292
  Male | 17 | 17 | 38 | 35 | 107
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 5 | 6 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 4 | 6 | 9 | 26
  White | 39 | 40 | 141 | 135 | 355
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 48 | 46 | 153 | 152 | 399

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity on Movement From 0-48 Hours Post-Treatment
Description: A derived measure computed based on a patient-reported numerical pain rating scale assessing pain as a whole number from 0 (no pain) to 10 (worst pain imaginable) when the subject sits up from a supine position. This measure was evaluated by electronic diary at 13 planned time points from 0 to 48 hours post-treatment. The values reported are mean pain scores for each treatment group.
Time Frame: Assessed from 0 to 48 hours post-dose, summary measure (see description) reported.
Population: mITT Population, results for only the prespecified analysis population {SABER-Bupivacaine (Part 2) and Bupivacaine HCl (Part 2)} are provided, there was no prespecified primary outcome measure that included the SABER-Bupivacaine (Part 1) arm or the Saline Placebo (Part 1) arm.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Part 2/SABER-Bupivacaine: 5 ml once at end of surgery
- Part 2/Bupivacaine HCl: 0.5%, 15 ml, once at end of surgery
Arm/Group | Part 2/SABER-Bupivacaine | Part 2/Bupivacaine HCl
Number analyzed (Participants) | 148 | 148
score on a scale | 5.55 (0.065) | 5.87 (0.059)
Statistical Analysis 1: Comparison: Part 2/SABER-Bupivacaine vs Part 2/Bupivacaine HCl; Pain Intensity on Movement 0-48 hr; Test type: Superiority — Primary; p = 0.124, ANOVA; Mixed model with repeated measures (MMRM) for scheduled pain measurements was estimated with time as a repeating factor within subject; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.84 to 0.10], Standard Error of Mean 0.24 — Least squares mean from the MMRM described in the Statistical Test of Hypothesis

2. Secondary Outcome: Pain Intensity Using the NPRS-11 With Movement
Description: A derived measure computed based on a patient-reported numerical pain rating scale assessing pain as a whole number from 0 (no pain) to 10 (worst pain imaginable) when the subject sits up from a supine position. This measure was evaluated by electronic diary at 17 planned time points from 0 to 72 hours post-treatment. The values reported are mean pain scores for each treatment group.
Time Frame: Assessed from 0 to 72 hours post-dose, summary measure (see description) reported.
Population: mITT Population, results for only the prespecified analysis population {SABER-Bupivacaine (Part 1 and Part 2 combined) and Bupivacaine HCl (Part 2)} are provided, there was no prespecified secondary outcome measure that included the Saline Placebo (Part 1) arm or the SABER-Bupivacaine (Part 1) arm as a standalone treatment group.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Part 1 and Part 2: SABER-Bupivacaine: 5 ml once at end of surgery
- Part 2: Bupivacaine HCl: 0.5%, 15 ml, once at end of surgery
Arm/Group | Part 1 and Part 2: SABER-Bupivacaine | Part 2: Bupivacaine HCl
Number analyzed (Participants) | 194 | 148
score on a scale | 4.94 (0.049) | 5.40 (0.052)

3. Secondary Outcome: Total IV Morphine-equivalent Dose of Rescue Opioids
Description: IV morphine-equivalent dose
Time Frame: 0-72 hrs. post dose (after surgery)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: IV morphine equivalent (mg)
Arm/Group | Part 1 and Part 2: SABER-Bupivacaine | Part 2: Bupivacaine HCl
Number analyzed (Participants) | 194 | 148
IV morphine equivalent (mg) | 21.4 (1.37) | 22.6 (1.58)

4. Secondary Outcome: Composite Endpoint of Silverman's Integrated Analgesic (SIA) Assessment Score
Description: Score of Integrated Analgesia (SIA) is a composite endpoint that integrates pain assessment scores with opioid use over various collections of timepoints by ranking the pain score and the opioid use separately across treatments. After the scores are computed the means are calculated across time points to provide a single overall treatment effect. The composite SIA score ranges from -200 to 200 with -200 being the best case and 200 the worst case.
Time Frame: 0 to 72 hours
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Part 1 and Part 2: SABER-Bupivacaine | Part 2: Bupivacaine HCl
Number analyzed (Participants) | 194 | 148
score on a scale | -17.3 (8.83) | -1.5 (9.33)

5. Secondary Outcome: Subjects Not Taking Rescue Medication From PACU Discharge to 72 Hours
Description: Pooled SABER-Bupivacaine parts 1 + 2 vs. Bupivacaine HCl
Time Frame: From PACU Discharge to 72 Hours post-treatment
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Part 1 and Part 2: SABER-Bupivacaine | Part 2: Bupivacaine HCl
Number analyzed (Participants) | 194 | 148
participants | 57 | 42

6. Secondary Outcome: Time to First Opioid Rescue Medication Use After Discharge From the PACU
Description: Pooled SABER-Bupivacaine parts 1 + 2 vs. Bupivacaine HCl
Time Frame: From PACU Discharge to 72 Hours post-treatment
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Part 1 and Part 2: SABER-Bupivacaine | Part 2: Bupivacaine HCl
Number analyzed (Participants) | 194 | 148
hours | 5.5 [3.5 to 7.7] | 6.1 [3.3 to 9.0]

7. Secondary Outcome: Time to PACU Discharge Eligibility as Assessed by Modified Post-Anesthesia Discharge Scoring System (mPADSS)
Description: mPADSS is a tool used to determine eligibility for discharge from the PACU after ambulatory surgery. It includes an assessment of parameters such as vital signs, activity level, nausea/vomiting, pain, and surgical bleeding. For this trial, evaluation of eligibility for PACU discharge by mPADSS has been slightly modified to provide a standardized means of assessing eligibility for PACU discharge across multiple investigative sites and also ensures that nonmedical complications, such as a missing ride home, do not interfere with evaluation of test drug effects.
Time Frame: From admission to discharge from PACU (Approximately 0 to 12 hours)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Part 1 and Part 2: SABER-Bupivacaine | Part 2: Bupivacaine HCl
Number analyzed (Participants) | 194 | 148
hours | 1.8 [1.8 to 1.9] | 1.9 [1.8 to 2.0]

ADVERSE EVENTS:
Time Frame: Approximately 0-60 days after surgery (duration of time over which each participant was assessed).
Description: Systematic and Non-systematic reported TEAEs of >5% (Safety Population)
Arm/Group | SABER-Bupivacaine (Part 1) | Saline Placebo (Part 1) | SABER-Bupivacaine (Part 2) | Bupivacaine HCL (Part 2)
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/47 | 0/148 | 0/148
Serious Adverse Events (participants affected / at risk) | 1/45 | 0/47 | 5/148 | 3/148
Other Adverse Events (participants affected / at risk) | 43/45 | 47/47 | 148/148 | 146/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SABER-Bupivacaine (Part 1) (N=45) | Saline Placebo (Part 1) (N=47) | SABER-Bupivacaine (Part 2) (N=148) | Bupivacaine HCL (Part 2) (N=148)
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SABER-Bupivacaine (Part 1) (N=45) | Saline Placebo (Part 1) (N=47) | SABER-Bupivacaine (Part 2) (N=148) | Bupivacaine HCL (Part 2) (N=148)
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 5 | 11
Constipation (Solicited) (Gastrointestinal disorders) | 20 | 19 | 65 | 58
Constipation (Gastrointestinal disorders) | 2 | 2 | 18 | 13
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 11 | 7
Dizziness (Nervous system disorders) | 1 | 2 | 13 | 14
Dizziness (Solicited) (Nervous system disorders) | 11 | 9 | 38 | 40
Dysgeusia (Solicited) (Gastrointestinal disorders) | 4 | 2 | 31 | 24
Dysgeusia (Nervous system disorders) | 1 | 0 | 13 | 9
Headache (Nervous system disorders) | 1 | 4 | 16 | 13
Headache (Solicited) (Nervous system disorders) | 17 | 15 | 53 | 49
Hypoaesthesia (Solicited) (Nervous system disorders) | 0 | 0 | 8 | 9
Incision site haemorrhage (Injury, poisoning and procedural complications) | 3 | 0 | 10 | 6
Incision site pain (Injury, poisoning and procedural complications) | 0 | 2 | 5 | 8
Nausea (Nervous system disorders) | 8 | 11 | 47 | 51
Nausea (solicited) (Nervous system disorders) | 10 | 15 | 42 | 45
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 5 | 2
Paraesthesia (Solicited) (Nervous system disorders) | 2 | 2 | 20 | 21
Post procedural contusion (Injury, poisoning and procedural complications) | 41 | 33 | 142 | 110
Post procedural discharge (Injury, poisoning and procedural complications) | 1 | 1 | 8 | 6
Procedural pain (Injury, poisoning and procedural complications) | 19 | 21 | 32 | 35
Pruritus (Solicited) (Skin and subcutaneous tissue disorders) | 5 | 11 | 31 | 27
Somnolence (Solicited) (Nervous system disorders) | 24 | 22 | 73 | 65
Somnolence (Nervous system disorders) | 1 | 0 | 16 | 12
Vomiting (Solicited) (Gastrointestinal disorders) | 7 | 7 | 10 | 17
vomiting (Gastrointestinal disorders) | 2 | 2 | 16 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/20/NCT02574520/Prot_SAP_000.pdf